CLINICAL TRIAL: NCT00535522
Title: A Multicenter, Open-Label, Noncomparative Phase I Clinical and Pharmacokinetic Study of Oral TAK-285 in Patients With Advanced Cancer
Brief Title: A Safety and Pharmacokinetic Study of TAK-285 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-285_101
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Cancer
Keywords: Pharmacokinetics; pharmacodynamics; maximal tolerated dose
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-285 (Experimental)
  Interventions: Drug: TAK-285 Dose Escalation Cohorts; Drug: TAK-285 Recommended Phase 2 Dosing Cohort

INTERVENTIONS:
Drug: TAK-285 Dose Escalation Cohorts — TAK-285 50 mg tablet, orally, once or twice daily for three weeks, followed by seven days off. Dose escalation to maximum tolerated dose, with possibility of continuous dosing per cycle (daily dosing for four weeks without a break between cycles).
Drug: TAK-285 Recommended Phase 2 Dosing Cohort — Expanded cohort with dose and regimen dependent upon the safety profile of the maximally tolerated dose and schedule determined in the dose escalation phase of the study.

SUMMARY:
The purpose of this study is to determine the safety and pharmacokinetics of TAK-285 in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria

* The subject has a histologically confirmed advanced non-hematologic malignancy.
* The subject has a chemotherapy-free interval of at least 4 weeks prior to first dose of study drug.
* The subject is intolerant of, is not a candidate for, or the subject's disease is refractory to established therapy known to provide clinical benefit for their disease.
* A female subject of childbearing potential who is sexually active agrees to use adequate contraception from Screening throughout the duration of the study, and for 30 days after the last dose of study drug. Male subjects should agree to use contraception for the duration of the study, and for 30 days after the last dose of study drug.
* The subject has a life expectancy of greater than 12 weeks.
* The subject has an Eastern Cooperative Oncology Group performance status of 0 to 2.
* The subject has the ability to swallow and retain oral medication
* The subject's most recent test values within 2 weeks before the date of entry meet the following standards:

  * Bone marrow function:

    * Absolute neutrophil count ≥1500/mm3
    * Hemoglobin ≥9.0g/dL, platelet count ≥100,000/mm3.
  * Liver function:

    * Total bilirubin ≤1.5 times the upper limit of the standard value of each institution
    * Aspartate aminotransferase and alanine aminotransferase ≤2.5 times the upper limit of the standard value of each institution.
  * Renal function:

    * Serum creatinine ≤1.5 times the upper limit of the standard value of each institution.
* In the recommended phase 2 dose Cohort, the subject has an accessible tumor for biopsy and is willing to undergo 2 tumor biopsies.
* In the recommended phase 2 dose Cohort, the subject has at least 1 measurable lesion based on the treatment assessment standards for solid tumors.
* In the recommended phase 2 dose Cohort, the subject has a tumor that expresses EGFR and/or overexpresses erbB2.

Exclusion Criteria

* The subject has a symptomatic brain metastasis.
* The subject has an uncontrollable pleural effusion, ascitic fluid, or pericardial effusion.
* The subject has active gastrointestinal bleeding as evidenced by either hematemesis or melena.
* The subject has acute gastrointestinal ulcers.
* The subject has been treated with a small molecule inhibitor of EGFR or HER2 (except for lapatinib).
* The subject has a history of any cancer other than the present condition (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 3 years.
* The subject has significant cardiovascular impairment (history of New York Heart Association class III or IV) or a history of myocardial infarction or unstable angina within the past 6 months prior to study drug treatment.
* The subject has a severe disease (other than cancer) that will likely affect the prospects of survival or a history that will make it difficult to appropriately manage and follow his or her progress in accordance with the protocol (serious organ disorder, mental illness, drug abuse, alcohol dependency, etc.).
* The subject requires prohibited treatment (drug, surgery or radiotherapy for treatment of malignant tumor, drugs that could interact with TAK-285) except for radiotherapy of limited area (<20% of total bone marrow) in order to relieve the symptoms from symptomatic bone metastasis.
* The subject who has been treated with a drug, which inhibits or induces Cytochrome P450 3A4 within 1 week prior to the start of treatment with the investigational drug.
* The subject is pregnant or breast feeding.
* The subject has participated in another clinical study/postmarketing clinical study within 4 weeks prior to the start of treatment with TAK-285.
* The subject is currently taking excluded medications, including:

  * Concurrent anticancer therapy with agents other than TAK-285.
  * The following prohibited medications and substances should not be used for at least 7 days prior to the start of the study and throughout completion:

    * Strong CYP3A4 inhibitors

      * Amiodarone
      * Diltiazem
      * Verapamil
      * Human immunodeficiency virus protease inhibitors
      * itraconazole
      * ketoconazole
      * macrolide antibiotics (excluding azithromycin)
    * Strong CYP3A4 inducers

      * Carbamazepine
      * Efavirenz
      * Nevirapine
      * Phenytoin
      * Rifabutin
      * Rifampin.
      * St. John's wort
    * Medications and devices containing hormones such as oral contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety profile, including dose-limiting toxicities, maximum tolerated dose, recommended Phase II dose; and the pharmacokinetic profile. | Duration of study

SECONDARY OUTCOMES:
Objective disease response by modified Response Evaluation Criteria in Solid Tumors. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Center, Detroit, Michigan

REFERENCES:
- [Derived] LoRusso P, Venkatakrishnan K, Chiorean EG, Noe D, Wu JT, Sankoh S, Corvez M, Sausville EA. Phase 1 dose-escalation, pharmacokinetic, and cerebrospinal fluid distribution study of TAK-285, an investigational inhibitor of EGFR and HER2. Invest New Drugs. 2014 Feb;32(1):160-70. doi: 10.1007/s10637-013-9988-x. Epub 2013 Jul 2. PMID 23817974